CLINICAL TRIAL: NCT06532448
Title: Evaluating the Feasibility of High-volume, Low-risk Penicillin Allergy De-labelling to Maximise Efficiency in a Resource-limited Setting
Acronym: De-Label Me
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RHM MED2073
Record Dates: First submitted 2024-07-29; First posted 2024-08-01 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-08

CONDITIONS: Penicillin Allergy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Single dose low-risk penicillin challenge — Initial screening to establish low risk allergy status followed by a single dose challenge using a standard penicillin dose. All challenges will be oral, conducted in a hospital setting and will be followed by a 1 hour monitoring period.

SUMMARY:
Plenty of studies have now established the safety of low-risk penicillin allergy de-labelling, but few have addressed how to organise de-labelling at the clinic level. This study will test the real world practicalities of running a de-labelling clinic optimised for maximum patient volume. The sheer number of patients with a penicillin allergy label, in contrast to relatively few allergy centres, makes demonstrating that such an approach can work extremely important for future antimicrobial stewardship.

DETAILED DESCRIPTION:
Participants with a penicillin allergy label will be invited to take part in the study, having been referred to the service by their hospital team. Based on the information provided with the referral, low-risk candidates will be identified.

Appointments will be offered to fill 36 clinic slots in total as part of the study.

On the day of their appointment, after providing written consent, participants will be asked some additional questions to confirm their eligibility for penicillin allergy de-labelling (and that the information provided in their referral form is accurate). Simple medical observations will also be taken (recording heart rate, blood pressure and oxygen saturation). Participants may be asked to return to the waiting area after these initial assessments.

Once a chair becomes available in the clinic, participants will be given a single dose of penicillin to take by mouth. They will then be observed for 1 hour. During this time they will be asked to complete a feedback form about their clinic experience.

Provided they do not experience a reaction they will then be discharged home, where they will be asked to complete a 3-day course of the same penicillin. They will be called during the next week to ensure that they completed the course and did not experience any delayed reactions. Their GP, and the person who referred to the service, will be informed of the outcome. Those that do not react will be able to receive penicillins in the future.

Participants should expect to be in the allergy department for up to 2 hours for their appointment.

The study does not need to be powered to make a specific statistical analysis possible; the intention is simply to demonstrate that a high-volume de-labelling service is viable. However, any one session may be affected by factors such as a high DNA rate, which would then mean that the clinic model is not tested at optimal capacity. To avoid this, and to make the overall results more compelling, the clinic will run on four occasions (with 36 patients in total).

ELIGIBILITY:
Inclusion Criteria:

1. Penicillin allergy label
2. Age ≥18
3. Registered as a patient with University Hospital Southampton NHS Foundation Trust (with a UHS medical record)
4. Able and willing to consent to penicillin de-labelling

Exclusion Criteria:

1. Penicillin allergy previously confirmed via positive blood, skin, BAT or challenge testing
2. PEN-FAST score >2 (indicating a moderate or high risk of a positive challenge)
3. Anaphylaxis, angioedema, wheeze, shortness of breath or suspected hypotension linked to treatment with penicillin
4. Received treatment in hospital for a reaction linked to penicillin (unless already an inpatient at onset)
5. Itchy or urticarial rash within 1 hour of starting a new course of treatment with penicillin
6. Severe cutaneous adverse reaction (SCAR) linked to penicillin exposure (e.g. SJS/TEN, DRESS), including symptoms suggestive of SCAR without a formal diagnosis (e.g. skin blistering or peeling, mucosal involvement)
7. History of other serious, non-immediate reactions linked to penicillin (e.g. haemolytic anaemia, transaminitis, nephritis)
8. Currently pregnant or breastfeeding
9. Poorly controlled asthma
10. Severe COPD
11. Severe or critical aortic stenosis
12. Clinically unstable secondary to other organ failure
13. Unwell or unstable on the day of proposed penicillin challenge (including acute febrile illness)
14. Prescribed other antibiotics on the day of proposed challenge, unless taken as a long-term treatment/prophylaxis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
How can low-risk penicillin allergy de-labelling be delivered with maximal efficiency in a resource limited setting? | 1 year
  Successful operation of the high-volume clinic model, assessed via:
  1. Number of patients reviewed and tested (if appropriate) within each allocated session
  2. Evidence of acceptability to patients from feedback forms

IPD SHARING:
Plan to Share IPD: No